CLINICAL TRIAL: NCT03041155
Title: Respiratory Muscle Training in Hemodialysis Patients: Effects on Physiologic Parameters and Endothelium-related Biomarkers
Brief Title: Respiratory Muscle Training in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Alexandre Braga Liborio, Visitant Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 43697715.0.0000.5054; NCT03075982 (obsolete NCT alias)
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): Muscle respiratory training
  Interventions: Behavioral: Muscle respiratory training
- control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Muscle respiratory training — Muscle respiratory training during hemodialysis sessions
  Arms: treatment

SUMMARY:
The research protocol is a Randomized Clinical Trial that has the effectiveness of a given respiratory muscle training protocol over the indicative variables: Pulmonary function; Markers of oxidative stress and inflammation, endothelial markers and Quality of life in patients with chronic kidney disease undergoing hemodialysis. According to the Investigators, this topic was proposed since it is known that several pulmonary complications occur as a consequence of chronic kidney disease due to uremic myopathy. Therefore, the hypothesis is that the application of a respiratory muscle training protocol will contribute positively pulmonary functionality and a decrease in oxidative stress and inflammation in chronic kidney patients, consequently, will bring improvement in the quality of life for these patients. The Patients will be divided into two groups: control group - No intervention of the Muscular Training (CG) And Intervention Group (GI). The intervention protocol will be composed of respiratory muscle training And lasts for two (2) months, with three (3) visits per week. It will be carried out through Threshold PeP appliance. The twelve (12) first training sessions will have a total duration of 30 minutes 15 minutes with inspiratory load of 20 cmH2O and 15 minutes with expiratory load of 20 CmH 2 O; and the others (12) twelve sessions will last 40 minutes each, with 20 minutes with an inspiratory load of 20 CmH2O and 20 minutes with expiratory load of 20 cmH2O. The variables evaluated will be: muscular strength Respiratory (maximum inspiratory pressure and maximum expiratory pressure - Pimáx and Pemáx); Lung function (Slow Vital Capacity - CVL, forced expiratory volume in the first minute - VEF1, Vital Capacity Forced - CVF and Maximum Voluntary Ventilation - VVM); Serum levels of oxidative stress markers, endothelial markers and endothelin.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis for more than 3 months
* No COPD diagnosis

Exclusion Criteria:

* Decompensated Heart failure
* Acute coronary disease in the last 3 months
* Active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
endothelium glycocalyx biomarkers | 8 weeks
  plasma syndecan-1 (ng/mL)

SECONDARY OUTCOMES:
Endothelium biomarker | 8 weeks
  ICAM (ng/mL)
Endotehlium Biomarker | 8 weeks
  VCAM(ng/mL)
Aberrant angiogenesis | 8 weeks
  Angiopoietin-2 (ng/mL)
Oxidative stress | 8 weeks
  Plasma Malondialdehyde (mmol/L)
Mean blood pressure | 8 weeks
  Blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Liborio, PHD, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Pronefron, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639